CLINICAL TRIAL: NCT03432806
Title: Development of Novel Imaging and Laboratory Biomarkers to Monitor the Liver Pre-metastatic Niche and Guide Treatment of Colon Cancer: A Pilot Study
Brief Title: A Study of Imaging, Blood, and Tissue Samples to Guide Treatment of Colon Cancer and Related Liver Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-594
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Liver Tumors
Keywords: Tissue samples; 17-594
MeSH Terms: conditions — Colonic Neoplasms; Carcinoma, Hepatocellular | interventions — Blood Specimen Collection; Colectomy; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- presumptive Stage II or III colon cancer
  Interventions: Other: blood draws; Procedure: colectomy or hepatectomy; Diagnostic Test: Fibroscan test
- Stage IV colon cancer with resectable hepatic metastases
  Interventions: Other: blood draws; Procedure: colectomy or hepatectomy; Diagnostic Test: Fibroscan test
- Stage IV colon cancer with unresectable hepatic metastases
  Interventions: Other: blood draws; Procedure: colectomy or hepatectomy; Diagnostic Test: Fibroscan test
- Stage I colon cancer, pre-neoplastic or benign colon lesions
  Interventions: Other: blood draws; Procedure: colectomy or hepatectomy

INTERVENTIONS:
Other: blood draws — Patients will have 10 mL of peripheral venous blood drawn immediately prior to surgery, in the post anesthesia care unit (PACU), and at the first postoperative clinic visit for a total of 30 mL.
Procedure: colectomy or hepatectomy — Three small pieces of otherwise "normal-appearing" liver of 0.5-1 cm3 collected intraoperatively from patients in all four groups (including Group D). Because liver biopsy is less frequently performed during operations for benign colon lesions or Stage I-III colon cancers, this single aspect of the protocol can be made optional at the discretion of the surgical attending or the patient, however bloods and tissue from pathology will still be collected.
Diagnostic Test: Fibroscan test — This may be done either at a preoperative clinic setting or immediately prior to surgery.
  Groups: Stage IV colon cancer with resectable hepatic metastases; Stage IV colon cancer with unresectable hepatic metastases; presumptive Stage II or III colon cancer

SUMMARY:
The purpose of this study is to explore novel ways of diagnosing colon cancer and predicting its propensity to spread to other organs such as the liver.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing one of the following procedures as part of their routine care in order to meet the inclusion criteria:

  * Operation for presumed stage I-IV colon cancer including colectomy, hepatectomy, or abdominal surgery (e.g. insertion of HAIP)
  * Colectomy for presumed benign or pre-malignant colon tumors (e.g. large nonneoplastic polyps or adenomas)
* Open, laparoscopic, or robotic resections
* ≥18 years old

Exclusion Criteria:

* Extrahepatic CRC metastasis
* No preoperative portal venous phase CT scan performed up to two months prior to day of surgery Pathology demonstrating a malignant tumor other than colorectal adenocarcinoma.
* Stage IV colon cancer with resectable hepatic disease undergoing hepatectomy with active primary colon tumor still in place (despite chemo-radiation therapy) and no plans for colectomy.
* Receipt of experimental therapies for colon cancer (e.g. checkpoint inhibitors or novel targeted agents). Of note, approved targeted agents (such as anti-angiogenic agents, EGFR inhibitors etc) are not an exclusion criterion.
* History of non-colonic malignancy w/in 5 years (except non-melanomatous skin cancer)
* Colon cancer with microsatellite instability (MSI-high) if known preoperatively
* Known hereditary colon cancer syndrome such as familial adenomatous polyposis (FAP) or hereditary nonpolyposis colorectal cancer (HNPCC)
* Known liver disease (e.g. non-alcoholic steatohepatitis, cirrhosis, viral or other form of hepatitis, etc)
* INR >2 or known clotting factor deficiency
* Anticipated need for full anticoagulation during hospitalization
* Receipt of medications that increase significantly the risk of bleeding after liver biopsy (at the surgeon"s discretion)
* Intraoperative discovery of pathology that precludes the planned surgical resection or liver biopsy, or makes resection futile (such as peritoneal carcinomatosis or other extrahepatic metastatic disease)
* Operating surgeon deems research interventions to be more than a minimal risk for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK clinic
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
successful isolation of exosomes | 1 year
  defined as isolation of at least 5μg of exosomal protein and reported as a binomial proportion with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Angelica, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm